CLINICAL TRIAL: NCT06837597
Title: Jianzhong Qushi Formula for Treating Chronic Radiation Induced Proctitis : a Multicenter, Prospective, Randomized Controlled Clinical Trial
Brief Title: Jianzhong Qushi in Chronic RRI
Acronym: ACRON
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Yirui Zhai,MD., Associate Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: No.24/520-4800
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Chronic Radiation Proctitis
Keywords: Chinese Tradiational Medicine; Chronic Radiation Proctitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Jianpi AnChang Group (Experimental): Jianzhong Qushi Formula, 100ml twice daily, taken before breakfast and after supper orally, for 28 days.
  Interventions: Drug: Jianzhong Qushi Formula
- Placebo Group (Placebo Comparator): Simulated Chinese medicine placebo, 100ml twice daily, taken before breakfast and after supper orally, for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Jianzhong Qushi Formula — Jianzhong Qushi Formula (A Chinese traditional formula, approved by Chinese Patent, No. ZL202210097886.0)
  Arms: Jianpi AnChang Group
Drug: Placebo — A simulated Chinese medicine placebo, with similar appearance and smell to Jianzhong Qushi Formula.
  Arms: Placebo Group

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled trial. Patients diagnosed as CRP and without TCM history will be enrolled and randomly assigned to either the treatment group (receiving standard care plus Jianzhong Qushi Formula, 100 ml bid, *28days) or the control group (receiving standard care plus placebo 100 ml bid, *28days). All of the patients received both The primary endpoint is the clinical response rate, defined as fulfilling one of the following, RTOG grade reduction, ① RTOG/EORTC grade reduction; ② ≥1 symptom downgraded by CTCAE v5.0; ③ Symptom improvement according to TCM symptom standards .The secondary endpoints included TCM syndrome score reduction rate, LENT/SOMA score changes, changes in gut microbiota, quality of life(QoL) , etc. Totally, 168 patients (84 in each group) will be enrolled.

DETAILED DESCRIPTION:
Both the treatment group and the control group are given standard treatment as recommended by the "2023 Edition of the Practice Guidelines for the Prevention and Treatment of Radiation Proctitis" or the "2018 Edition of the Expert Consensus on the Diagnosis and Treatment of Radiation Proctitis in China", such as sucralfate/steroids/loperamide according to symptoms.

① Treatment Group: Administer Jianzhong Qushi Formula, 100ml per dose, twice daily, taken before breakfast and after dinner, for a total of 28 days.

② Control Group: Administer a simulated Chinese medicine placebo, 100ml per dose, twice daily, taken before breakfast and after dinner, for a total of 28 days.

Observational medication

Jianzhong Qushi Formula (Patent No.: ZL202210097886.0) Composition:

* Monarch medicines (jun yao): Codonopsis (Dang Shen) tonifies the spleen and strengthens the body, serving as the monarch medicine.

  * Minister medicines (chen yao): Atractylodes Macrocephala (Bai Zhu) is heavily used to dry dampness, transform phlegm, strengthen the spleen, and boost energy, along with Pinellia (Ban Xia) which is good at descending adverse qi and stopping vomiting, drying dampness and strengthening the spleen; both serve as the minister medicines.

    * Assistant medicines (zuo yao): Poria (Fu Ling), Tangerine Peel (Chen Pi), and Amomum Tsao-ko (Cao Guo): serve to promote diuresis and reduce dampness to stop diarrhea, regulate qi to relieve abdominal pain, and dry dampness to resolve phlegm; Syzygium aromaticum (Ding Xiang) and Magnolia Officinalis (Hou Po) regulate qi and strengthen the spleen, Aucklandia Lappa (Mu Xiang) has a fragrant aroma that dries dampness, awakens the spleen, and harmonizes the middle burner, also assisting Amomum Tsao-ko and Tangerine Peel in drying dampness and resolving phlegm; Aspergillus Oryzae (Shen Qu) enters the spleen and stomach meridians, has the function of promoting digestion and appetite, and also regulates qi and resolves dampness, harmonizing the spleen and stomach; Codonopsis Pilosula (Bai Lian) regulates qi; Taraxacum Mongolicum (Pu Gong Ying) and Bletilla Stripping (Bai Ji) are combined to clear heat and detoxify, reduce swelling and disperse blood stasis, detoxify and resolve blood stasis obstruction, all serving as the assistant medicines.

      * Guide medicines(shi yao): Glycyrrhiza Uralensis (Zhi Gan Cao) harmonizes all the medicines and serves as the guide medicines.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 years old
* ECOG score ≤ 2
* Pathologically confirmed malignant tumor
* Received pelvic radiotherapy, and it has been ≥ 3 months since the end of radiotherapy ;
* Meet the diagnostic criteria for chronic radiation proctitis in the "2023 Edition of the Practice Guidelines for the Prevention and Treatment of Radiation Proctitis" or the "2023 Edition of the Expert Consensus on the Diagnosis and Treatment of Radiation Intestinal Injury in Traditional Chinese and Western Medicine in China", with an international grading of level 1 - 2
* Meet the syndrome of spleen deficiency , and the syndrome differentiation is determined according to the "2017 Edition of the Expert Consensus on the Diagnosis and Treatment of Radiation Proctitis (Intestinal Syndrome) in Traditional Chinese Medicine" formulated by the Oncology Branch of the China Association of Traditional Chinese Medicine : Basic Syndrome PRO Scale of Spleen Deficiency (meeting 2 main symptoms or 1 main symptom* + 2 secondary symptoms#).
* Hemoglobin ≥ 100 g / L, neutrophils ≥ 1.5 × 10^9^ / L
* Serum creatinine ≤ 1.25 times the upper normal limit (UNL)
* Total bilirubin ≤ 1.5 times UNL, alanine aminotransferase and aspartate aminotransferase ≤ 2.5 times UNL
* The patient has signed the informed consent form
* The patient agrees to cooperate with the follow - up. *Main symptoms included abdominal distension ,anorexia,tenesmus, unsatisfactory bowel movement and fatigue.

  * Secondary symptoms included spontaneous sweating, dizziness,feeling of heaviness in the head, feeling of heaviness in the body, nausea and palpitations.

Exclusion Criteria:

* Other causes of enteritis cannot be ruled out
* The relevant symptoms existed before radiotherapy and did not worsen after treatment
* Allergy to more than 3 components of the Western medicine used in this study or the formula of Jianzhong Qushi Formula
* Tumor progression requiring urgent anti-tumor treatment
* Urgent surgical or endoscopic treatment is needed
* Has already entered other clinical studies targeting RRI
* Nursing or pregnant women
* Those who may interfere with the study evaluation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Response rate | 1-month, 3-month, 6-month
  ① A downgrade in the RTOG/EORTC radiation proctitis grading; ② A downgrade in the evaluation of ≥1 radiation enteritis - related symptom according to the National Cancer Center of the United States Common Terminology Criteria for Adverse Events 5.0 (CTCAE 5.0 ); ③ Syndrome: alleviation of 2 main symptoms or 1 main symptom + 2 secondary symptoms

SECONDARY OUTCOMES:
Change of TCM syndrome scores: Calculated as (Pre-treatment Syndrome Score - Post-treatment Syndrome Score) / Pre-treatment Syndrome Score×100%. (Refer to the relevant standards in the "Guiding Principles for Clinical Research on New Traditional | 1-month, 3-month, 6-month
  Higher means better
Changes in Late Effects Normal Tissue Task Force (LENT)-Subjective, Objective, Management, Analytic (SOMA) scales | 1-month, 3-month, 6-month
  Fewer score means better
Changes in Quality of Life Scores | 1-month, 3-month, 6-month
  Higher score means better
Changes in intestinal flora | 1-month, 3-month, 6-month

CONTACTS AND LOCATIONS:
Overall Officials: Li Feng, MD., Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing may be limited by agreements with sponsors, collaborators, or regulatory bodies, as well as jurisdictional laws governing data protection , for academic use only (non-commercial, non-political).

REFERENCES:
- [Background] Tabaja L, Sidani SM. Management of Radiation Proctitis. Dig Dis Sci. 2018 Sep;63(9):2180-2188. doi: 10.1007/s10620-018-5163-8. PMID 29948565
- [Background] Denton A, Forbes A, Andreyev J, Maher EJ. Non surgical interventions for late radiation proctitis in patients who have received radical radiotherapy to the pelvis. Cochrane Database Syst Rev. 2002;(1):CD003455. doi: 10.1002/14651858.CD003455. PMID 11869662
- [Background] Liu L, Xiao N, Liang J. Comparative efficacy of oral drugs for chronic radiation proctitis - a systematic review. Syst Rev. 2023 Aug 22;12(1):146. doi: 10.1186/s13643-023-02294-2. PMID 37608385
- [Background] Sahebnasagh A, Ghasemi A, Akbari J, Alipour A, Lashkardoost H, Ala S, Hosseinimehr SJ, Salehifar E. Prevention of acute radiation-induced Proctitis by Aloe vera: a prospective randomized, double-blind, placebo controlled clinical trial in Pelvic Cancer patients. BMC Complement Med Ther. 2020 May 13;20(1):146. doi: 10.1186/s12906-020-02935-2. PMID 32404169
- [Background] Vanneste BG, Van De Voorde L, de Ridder RJ, Van Limbergen EJ, Lambin P, van Lin EN. Chronic radiation proctitis: tricks to prevent and treat. Int J Colorectal Dis. 2015 Oct;30(10):1293-303. doi: 10.1007/s00384-015-2289-4. Epub 2015 Jul 23. PMID 26198994
- [Background] Clarke RE, Tenorio LM, Hussey JR, Toklu AS, Cone DL, Hinojosa JG, Desai SP, Dominguez Parra L, Rodrigues SD, Long RJ, Walker MB. Hyperbaric oxygen treatment of chronic refractory radiation proctitis: a randomized and controlled double-blind crossover trial with long-term follow-up. Int J Radiat Oncol Biol Phys. 2008 Sep 1;72(1):134-143. doi: 10.1016/j.ijrobp.2007.12.048. Epub 2008 Mar 14. PMID 18342453